CLINICAL TRIAL: NCT02605837
Title: Oral Budesonide Suspension (OBS) in Adolescent and Adult Subjects (11 to 55 Years of Age, Inclusive) With Eosinophilic Esophagitis: A Phase 3 Randomized, Double-blind, Placebo-controlled Study
Brief Title: A Study in Adolescents and Adults With Eosinophilic Esophagitis (EoE) Measuring Histologic Response and Determine if Reduction in Dysphagia is Achieved
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHP621-301
Record Dates: First submitted 2015-11-04; First posted 2015-11-16 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2021-05

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Budesonide Suspension (OBS) (Experimental): Participants will receive Oral Budesonide Suspension (OBS) 10 milliliter (ml) of 0.2 milligram per milliliter (mg/ml) twice daily up to 16 weeks.
  Interventions: Drug: Oral Budesonide Suspension (OBS)
- Placebo (Placebo Comparator): Participants will receive oral dose of 10 ml of placebo matched with the experimental drug twice daily up to 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Budesonide Suspension (OBS) — Oral Budesonide Suspension (OBS) 10 milliliter (ml) of 0.2 milligram per milliliter (mg/ml) twice daily up to 16 weeks.
  Arms: Oral Budesonide Suspension (OBS)
Drug: Placebo — Oral dose of 10 ml of placebo matched with the experimental drug.
  Arms: Placebo

SUMMARY:
A study in adolescents and adults with eosinophilic esophagitis (EoE) to measure the histologic response and determine if any reduction in dysphagia is achieved.

ELIGIBILITY:
Inclusion Criteria

* Participants is able to provide written informed consent (participant, parent or legal guardian, and, as appropriate, participant assent) to participate in the study before completing any study-related procedures.
* Participant is male or female aged 11-55 years, inclusive, at time of consent.
* Participant has histologic evidence of eosinophilic esophagitis (EoE) with a peak eosinophil count of greater than or equal to (>=) 15/ high-powered field (HPF), from 2 of 3 (proximal, mid-, and/or distal) levels of the esophagus at the screening endoscopy.
* Participant has a history of clinical symptoms of esophageal dysfunction (for example, eating problems, abdominal pain, heartburn, dysphagia, vomiting, food impaction, weight loss) intermittently or continuously at screening (Visit -1).
* Participants must have experienced dysphagia (response of "yes" to question 2 on Dysphagia Symptom Questionnaire [DSQ]) on a minimum of 4 days and completed the DSQ on >= 70 percent (%) of days in any 2 consecutive weeks of the screening period and in the last 2 weeks prior to the baseline visit (Visit 1).
* Participant must not have PPI-responsive EoE based on esophageal biopsies performed after the patient has been on at least 8 weeks of high-dose PPI therapy (high-dose therapy refers to the total daily dose, which may have been administered as a once or twice daily dosing regimen). This may occur at the time of the qualifying esophagogastroduodenoscopy (EGD) (in which case the same proton pump inhibitor (PPI) regimen must be continued), or this may have been done previously (in which case PPI therapy may have been stopped if there was no response to therapy based on esophageal biopsy results). If PPI responsiveness was excluded by a previous EGD and biopsy, the historical EGD and biopsy must have been performed after the patient had been on a minimum of 6 weeks of high-dose PPI therapy.
* Participant will be on a stable (no changes) diet >=3 months prior to the screening visit (Visit -1).
* Participant is willing and able to continue any dietary therapy, environmental therapy, and/or medical regimens (including gastric acid suppression) in effect at the screening visit (Visit -1). There should be no change to these regimens during study participation.
* All female participants must have a negative serum pregnancy test (beta-human chorionic gonadotropin [β-hCG]) prior to enrollment into the study. Females of childbearing potential must agree to continue acceptable birth control measures (for example, abstinence, stable oral contraceptives, or double-barrier methods) throughout study participation.
* Participant is willing and has an understanding and ability to fully comply with study procedures and restrictions defined in this protocol.

Exclusion Criteria

* Participant has any condition or abnormality (including laboratory abnormalities), current or past, that, in the opinion of the principal investigator or medical monitor, would compromise the safety of the participant or interfere with or complicate the assessment of signs or symptoms of EoE. Such conditions may include psychiatric problems; neurologic deficits or disease; developmental delay; cardiovascular, metabolic, or pulmonary disease; or previous gastroesophageal surgery. These should be discussed with the medical monitor.
* Participant has used immunomodulatory therapy within 8 weeks prior to the qualifying EGD or between the qualifying EGD and baseline visit (Visit 1) or anticipates using immunomodulatory therapy during the treatment period (except for any ongoing regimen of allergy shots). Use of long-acting immunomodulatory therapy (for example, Rituxan) within 3 months of the qualifying EGD should be reviewed with the medical monitor.
* Participant has been using swallowed topical corticosteroid for EoE or systemic corticosteroid for any condition within the 4 weeks prior to the qualifying EGD, between the qualifying EGD and baseline visit (Visit 1), or anticipates use during the treatment period; any temporary use (less than or equal to [<=]7 days) or initiation of new steroid treatment during the study should be documented and discussed with the medical monitor prospectively but cannot occur within 4 weeks of the final EGD.
* Participant has been on inhaled steroids and has not been on stable treatment for >=3 months prior to screening visit (Visit -1). Participants on inhaled steroids need to stay on a stable treatment during study participation. Participant has been on intranasal steroids and has not been on stable treatment for a minimum of 4 weeks prior to the qualifying EGD. After the qualifying EGD, participants with seasonal allergic rhinitis may resume (or discontinue) intranasal corticosteroids based on the participant's usual treatment regimen for allergy season.
* Participant has initiated, discontinued, or changed dosage regimen of PPIs, H2 antagonists, antacids, or leukotriene inhibitors for any condition (such as gastroesophageal reflux disease, asthma or allergic rhinitis) within the 4 weeks prior to the qualifying EGD, between the qualifying EGD and baseline visit (Visit 1), or anticipates changes in the use of such medications during the treatment period.
* Participant has been using cytochrome P450 3A4 (CYP450 3A4) inhibitors (for example, ketoconazole, grapefruit juice) within the 2 weeks prior to the baseline visit (Visit 1) or within 5 half-lives (whichever is greater) or anticipates using such medications during the treatment period.
* Participant has an appearance on qualifying EGD of an esophageal stricture (high-grade), as defined by the presence of a lesion that does not allow passage of a diagnostic adult upper endoscope (for example, with an insertion tube diameter of greater than [>]9 millimeter [mm]).
* Participant is on a pure liquid diet or the 6-food elimination diet.
* Participant has had an esophageal dilation within the 3 months prior to screening (Visit -1).
* Participant has presence of esophageal varices at the screening endoscopy.
* Participant has any current disease of the gastrointestinal tract, aside from EoE, including eosinophilic gastritis, enteritis, colitis, or proctitis; inflammatory bowel disease; or celiac disease.
* Participant has other diseases causing or associated with EoE, including hypereosinophilic syndrome, collagen vascular disease, vasculitis, achalasia, or parasitic infection.
* Participant has current evidence of oropharyngeal or esophageal candidiasis.
* Participant has a potentially serious acute or chronic viral infection or immunodeficiency condition, including tuberculosis, fungal, bacterial, viral/parasite infection, ocular herpes simplex, herpes esophagitis, or chicken pox/measles.
* Participant has upper gastrointestinal bleeding within 4 weeks prior to the screening visit (Visit - 1) or between the screening visit and baseline visit (Visit 1).
* Participant has evidence of active infection with Helicobacter pylori.
* Participant has evidence of unstable asthma within 4 weeks prior to the screening visit (Visit -1) and between the screening visit and baseline visit (Visit 1).
* Participant is female and pregnant or nursing.
* Participant has a history of intolerance, hypersensitivity, or idiosyncratic reaction to budesonide (or any other corticosteroids) or to any other ingredients of the investigational product.
* Participant has taken part and received intervention in an interventional study related to EoE (except for an interventional study for a topical swallowed steroid) within 6 months prior to the screening visit (Visit -1), or any investigational study within 30 days prior to the screening visit (Visit -1). An investigational topical swallowed steroid must have been discontinued at least 30 days prior to the screening visit (Visit -1).
* Participant has a history or high risk of noncompliance with treatment or regular clinic visits.
* Participant has previously completed, discontinued, or withdrawn from this study.
* Participant has participated in a previous clinical study involving oral budesonide suspension (OBS) (SHP621).
* Participant anticipates using sucralfate during the study.

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 318 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (76):
- United States (76):
  - Children's Hospital, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Del Sol Research Management, Tucson, Arizona
  - Adobe Clinical Research LLC, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - GW Research, Inc., Chula Vista, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Colorado Children's Hospital, Aurora, Colorado
  - Asthma and Allergy Associates PC, Colorado Springs, Colorado
  - Rocky Mountain Pediatric Gastroenterology, Lone Tree, Colorado
  - Rocky Mountain Clinical Research LLC, Wheat Ridge, Colorado
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Connecticut GI, PC - Research Division, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nature Coast Clinical Research LLC, Inverness, Florida
  - Borland Groover Clinic, Jacksonville, Florida
  - Arnold Palmer Hospital For Children, Orlando, Florida
  - Accord Clinical Research LLC, Port Orange, Florida
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Center for Children's Digestive Health, Park Ridge, Illinois
  - University of Illinois College of Medicine at Peoria Pediatric Subspecialty Clinic, Peoria, Illinois
  - OSF St Francis Medical Center, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - Gastroenterology of Southern Indiana, New Albany, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Gastroenterology Associates LLC, Baton Rouge, Louisiana
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - Clinical Trials of America LA LLC - PPDS, West Monroe, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - West Michigan Clinical Research, Wyoming, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Minnesota Gastroenterology PA, Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - South Jersey Gastroenterology, Marlton, New Jersey
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - Mount Sinai Hospital, New York, New York
  - Asheville Gastroenterology Associates PA, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Clinical Trials of America-NC, LLC - PPDS, Mount Airy, North Carolina
  - Consultants For Clinical Research Inc, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Gastrointestinal and Liver Diseases Consultants PC, Dayton, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Endoscopy and Research Center, Houston, Texas
  - Digestive Health Center, Pasadena, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Advanced Research Institute, Ogden, Utah
  - Primary Children's Hospital, University of Utah, Salt Lake City, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Emeritas Research Group, Lansdowne Town Center, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- [Derived] Dellon ES, Collins MH, Katzka DA, Mukkada VA, Falk GW, Zhang W, Goodwin B, Terreri B, Boules M, Desai NK, Hirano I. Effect of randomized treatment withdrawal of budesonide oral suspension on clinically relevant efficacy outcomes in patients with eosinophilic esophagitis: a post hoc analysis. Therap Adv Gastroenterol. 2024 Dec 23;17:17562848241307602. doi: 10.1177/17562848241307602. eCollection 2024. PMID 39735351
- [Derived] Hirano I, Collins MH, Katzka DA, Mukkada VA, Falk GW, Terreri B, Boules M, Zhang W, Desai NK, Dellon ES. Effect of Esophageal Dilation History on Efficacy Outcomes in Patients With Eosinophilic Esophagitis Receiving Budesonide Oral Suspension. Am J Gastroenterol. 2024 Nov 12;120(7):1502-1510. doi: 10.14309/ajg.0000000000003197. PMID 39631042
- [Derived] Mukkada VA, Gupta SK, Gold BD, Dellon ES, Collins MH, Katzka DA, Falk GW, Williams J, Zhang W, Boules M, Hirano I, Desai NK. Pooled Phase 2 and 3 Efficacy and Safety Data on Budesonide Oral Suspension in Adolescents with Eosinophilic Esophagitis. J Pediatr Gastroenterol Nutr. 2023 Dec 1;77(6):760-768. doi: 10.1097/MPG.0000000000003948. Epub 2023 Sep 18. PMID 37718471
- [Derived] Dellon ES, Collins MH, Katzka DA, Mukkada VA, Falk GW, Morey R, Goodwin B, Eisner JD, Lan L, Desai NK, Williams J, Hirano I; ORBIT2/SHP621-302 Investigators. Long-Term Treatment of Eosinophilic Esophagitis With Budesonide Oral Suspension. Clin Gastroenterol Hepatol. 2022 Jul;20(7):1488-1498.e11. doi: 10.1016/j.cgh.2021.06.020. Epub 2021 Jun 26. PMID 34182150
- [Derived] Hirano I, Collins MH, Katzka DA, Mukkada VA, Falk GW, Morey R, Desai NK, Lan L, Williams J, Dellon ES; ORBIT1/SHP621-301 Investigators. Budesonide Oral Suspension Improves Outcomes in Patients With Eosinophilic Esophagitis: Results from a Phase 3 Trial. Clin Gastroenterol Hepatol. 2022 Mar;20(3):525-534.e10. doi: 10.1016/j.cgh.2021.04.022. Epub 2021 Apr 19. PMID 33887475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 72 sites in North America from 07 December 2015 (first participant enrolled) to 15 February 2019 (last participant completed).
Pre-assignment Details: A total of 318 participants were randomized and received the treatment (placebo or oral Budesonide suspension [OBS]) in a double blind fashion following a placebo lead-in phase and 296 participants completed the study.
Groups:
- Placebo: Participants received oral dose of 10 milliliter (ml) placebo matched with the Oral Budesonide Suspension (OBS) twice daily up to 16 weeks.
- Oral Budesonide Suspension (OBS): Post placebo lead in phase (4 weeks) participants received OBS 10 ml (2 mg) twice daily up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Started | 105 | 213
Completed | 94 | 202
Not Completed | 11 | 11
Not completed — Adverse Event | 3 | 1
Not completed — Non-Compliance with Study Drug | 0 | 1
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received at least one dose of a double-blind investigational product (IP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Oral Budesonide Suspension (OBS) | Total
Number analyzed (Participants) | 105 | 213 | 318
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age was calculated as the difference between date of birth and date of informed consent, truncated to years.
  Years | 33.9 (12.13) | 33.8 (11.89) | 33.9 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 84 | 127
  Male | 62 | 129 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 10
  Not Hispanic or Latino | 100 | 204 | 304
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 5 | 5
  White | 101 | 200 | 301
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Histologic Response at the Final Treatment Period Evaluation (Week 16)
Description: Histologic response was defined as a peak eosinophil count of less than or equal to (<=) 6/ high-powered field (HPF) across all available esophageal levels at final treatment period evaluation (Week 16). Histologic response after 12 weeks of double blind treatment at Week 16 was reported.
Time Frame: Week 16
Population: FAS included all randomized participants who received at least one dose of a double-blind IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 105 | 213
Participants
  Histology Response - Yes | 1 | 113
  Histology Response - No | 104 | 100
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); The Cochran-Mantel-Haenszel (CMH) adjusted difference in proportion with corresponding Newcombe confidence interval (CI) and odds ratio with corresponding CI were based on CMH test stratified by age group and diet restriction; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportion of responders = 0.52, 95% CI [0.433 to 0.591]

2. Primary Outcome: Number of Participants With Dysphagia Symptom Response at the Final Treatment Period Evaluation (Week 16)
Description: Dysphagia symptom response was defined as greater than or equal to (>=) 30 percent (%) reduction in the Dysphagia Symptom Questionnaire (DSQ) combined score (questions 2+3). DSQ contained 4 questions, all participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). DSQ score= ([sum of points from questions 2+3 in the daily DSQ]×14)/ Number of diaries reported with non-missing data. Dysphagia symptom response after 12 weeks of double blind treatment at Week 16 was reported.
Time Frame: Week 16
Population: FAS included all randomized participants who received at least one dose of a double-blind IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 105 | 213
Participants
  Dysphagia symptom response: Yes | 41 | 112
  Dysphagia symptom response: No | 64 | 101
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); The CMH adjusted difference in proportion with corresponding Newcombe confidence interval (CI) and odds ratio with corresponding CI were based on CMH test stratified by age group and diet restriction; Test type: Superiority; p = 0.024, Cochran-Mantel-Haenszel; Difference in proportion of responders = 0.13, 95% CI [0.016 to 0.243]

3. Secondary Outcome: Change From Baseline in Dysphagia Symptom Questionnaire (DSQ) Combined Score at the Final Treatment Period Evaluation (Week 16)
Description: DSQ contained 4 questions, all participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). DSQ combined score= ([sum of points from questions 2+3 in the daily DSQ]×14)/ Number of diaries reported with non-missing data. Scale range was 0 - 2 for question 2 and 0 - 4 for question 3, with higher values representing a worse outcome. Scale range for DSQ combined score was 0 - 84, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased. Change from baseline in DSQ after 12 weeks of double blind treatment at Week 16 was reported.
Time Frame: Baseline, Week 16
Population: FAS included all randomized participants who received at least one dose of a double-blind IP. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 89 | 197
Score on scale | -9.07 (1.519) | -12.99 (1.202)
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); This analysis was from analysis of covariance (ANCOVA) model with treatment group and age group as factors and the baseline DSQ combined score as a continuous covariate; Test type: Superiority; p = 0.015, ANCOVA; Difference in Least square mean = -3.92, 95% CI [-7.073 to -0.774]

4. Secondary Outcome: Change From Baseline in Total Endoscopy Score at the Final Treatment Period Evaluation (Week 16)
Description: Endoscopic findings with separate evaluations of the proximal and distal esophagus were recorded with respect to 5 categories: 1) exudates or plaques (grade 0-2); 2) fixed esophageal rings (grade 0-3); 3) edema (grade 0-2); 4) furrows (grade 0-2); and 5) strictures (grade 0-1). An endoscopy score for each category was calculated and summed for each anatomic location (proximal and distal). The minimum and maximum endoscopy score was 0 and 10 points respectively for each location (proximal and distal) and the total endoscopy score was the sum of the scores for the proximal and distal locations (maximum total score of 20 points respectively). The higher score indicated worse appearance. A negative change from baseline indicates that appearance improved. Endoscopic findings after 12 weeks of double blind treatment at Week 16 were reported.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 93 | 202
score on scale | -2.2 (0.38) | -4.0 (0.30)
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); This analysis was from analysis of covariance (ANCOVA) model with treatment group and age group as factors and the baseline. Total EREFS (endoscopy score) as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; Difference in Least square mean = -1.8, 95% CI [-2.6 to -1.1]

5. Secondary Outcome: Number of Participants With Peak Eosinophil Count Less Than (<)15/High-Powered Field (HPF) or Less Than or Equal to (<=)1/High-Powered Field (HPF) at the Final Treatment Period Evaluation (Week 16)
Description: Participant was considered as responder at Week 16 if he/she had peak eosinophil count of <15/HPF or <=1/HPF across all esophagus levels. Number of participants with peak eosinophil count < 15/HPF or <=1/HPF after 12 weeks of double blind treatment at Week 16 were reported.
Time Frame: Week 16
Population: FAS included all randomized participants who received at least one dose of a double-blind IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 105 | 213
Participants
  Peak Eosinophil Count (<15/HPF): Responders | 1 | 132
  Peak Eosinophil Count (<15/HPF): Non-responders | 104 | 81
  Peak Eosinophil Count (<=1/HPF): Responders | 0 | 69
  Peak Eosinophil Count (<=1/HPF): Non-responders | 105 | 144
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); Peak eosinophil count (<15/HPF) was performed based on logistic regression model adjusted for age group and diet restriction; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 169.74, 95% CI [23.235 to 1239.979]
Statistical Analysis 2: Comparison: Placebo vs Oral Budesonide Suspension (OBS); Peak eosinophil count (<=1/HPF) was performed based on firth logistic regression model adjusted for age group and diet restriction; Test type: Superiority; p = 0.001, Firth logistic regression; Odds Ratio (OR) = 100.69, 95% CI 2-sided [6.294 to 1610.749]

6. Secondary Outcome: Change From Baseline in the Peak Eosinophil Count at the Final Treatment Period Evaluation (Week 16)
Description: Change from baseline in the peak eosinophil count after 12 weeks of double blind treatment at week 16 for each available esophageal level (proximal, mid, distal, maximum) were reported.
Time Frame: Baseline, Week 16
Population: FAS included all randomized participants who received at least one dose of a double-blind IP. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure at each specific category.
Measure: Least Squares Mean (Standard Error); unit: eosinophil count
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 105 | 213
eosinophil count
  Proximal: Week 16: number analyzed (Participants) | 92 | 201
  Proximal: Week 16 | -5.5 (3.19) | -34.0 (2.52)
  Mid: week 16: number analyzed (Participants) | 92 | 199
  Mid: week 16 | -12.9 (3.74) | -43.3 (3.01)
  Distal: Week 16: number analyzed (Participants) | 91 | 201
  Distal: Week 16 | -4.9 (3.66) | -38.0 (2.88)
  Maximum: Week 16: number analyzed (Participants) | 92 | 201
  Maximum: Week 16 | -7.6 (4.27) | -55.2 (3.37)
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); This analysis of proximal eosinophil count was from the analysis of covariance (ANCOVA) model with treatment group and age group as factors and the baseline Peak Eosinophil Count as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; Difference in Least square mean = -28.4, 95% CI [-35.0 to -21.8]
Statistical Analysis 2: Comparison: Placebo vs Oral Budesonide Suspension (OBS); This analysis of mid eosinophil count was from the analysis of covariance (ANCOVA) model with treatment group and age group as factors and the baseline Peak Eosinophil Count as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; Difference in Least square mean = -30.4, 95% CI [-38.1 to -22.7]
Statistical Analysis 3: Comparison: Placebo vs Oral Budesonide Suspension (OBS); This analysis of distal eosinophil count was from the analysis of covariance (ANCOVA) model with treatment group and age group as factors and the baseline Peak Eosinophil Count as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; Difference in Least square mean = -33.1, 95% CI [-40.7 to -25.5]
Statistical Analysis 4: Comparison: Placebo vs Oral Budesonide Suspension (OBS); This analysis of maximum eosinophil count was from the ANCOVA model with treatment group and age group as factors and the baseline Peak eosinophil count as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Mean = -47.6, 95% CI 2-sided [-56.4 to -38.8]

7. Secondary Outcome: Change From Baseline in the Histopathologic Epithelial Features Combined Total Score Ratio (TSR) at the Final Treatment Period Evaluation (Week 16)
Description: Change from baseline in histopathologic epithelial features combined total score of grade and stage ratio after 12 weeks of double blind treatment at Week 16 were reported by measuring eight histopathologic epithelial features: basal layer hyperplasia, eosinophil density, eosinophil micro-abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells, lamina propria fibrosis were scored on a 4-point scale (0=normal, 3=worst) for both the severity of the abnormality (grade) and the amount of tissue affected by the abnormality (stage). Thus each of the 3 levels had a minimum score of 0 and maximum possible score of 24, and a possible total grade or stage score of 72 for a maximum combined score of 144. Combined total score ratio (TSR) =(proximal TSR + mid TSR + distal TSR)/N, where N is the number of non missing sections for TSR. A negative change from baseline indicates that epithelial inflammation decreased.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 92 | 201
score on scale
  Grade - Combined TSR: Week 16 | -0.03 (0.016) | -0.22 (0.013)
  Stage - Combined TSR: Week 16 | -0.0 (0.02) | -0.2 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); This analysis of histopathologic epithelial features combined grade TSR was from the analysis of covariance (ANCOVA) model with treatment group and age group as factors and the baseline Peak Eosinophil Count as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; Difference in Least square mean = -0.19, 95% CI [-0.22 to -0.16]
Statistical Analysis 2: Comparison: Placebo vs Oral Budesonide Suspension (OBS); This analysis of histopathologic epithelial features combined stage TSR was from the analysis of covariance (ANCOVA) model with treatment group and age group as factors and the baseline Peak Eosinophil Count as a continuous covariate; Test type: Superiority; p < 0.001, ANCOVA; Difference in Least square mean = -0.2, 95% CI [-0.2 to -0.2]

8. Secondary Outcome: Number of Participants With Dysphagia Symptom Response (Binary Response) at the Final Treatment Period Evaluation (Week 16)
Description: Dysphagia symptom response (binary response [i.e, responders versus. non-responders]) was defined as a >=50% reduction in the DSQ combined score (questions 2+3), from baseline to the final treatment period evaluation (Week 16). DSQ contained 4 questions, all participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). DSQ score= ([sum of points from questions 2+3 in the daily DSQ]×14)/ Number of diaries reported with non-missing data. Number of participants with binary response after 12 weeks of double blind treatment at Week 16 were reported.
Time Frame: Week 16
Population: FAS included all randomized participants who received at least one dose of a double-blind IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 105 | 213
Participants
  Responders | 35 | 88
  Non Responders | 70 | 125
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); Dysphagia symptom response (binary response) at the final treatment period was performed based on logistic regression model adjusted for age group and diet restriction; Test type: Superiority; p = 0.164, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.866 to 2.333]

9. Secondary Outcome: Number of Participants With Overall Binary Response I at the Final Treatment Period Evaluation (Week 16)
Description: Overall binary response I was defined as a reduction in the DSQ score of >=30% from baseline to the final treatment period (week 16) evaluation and a peak eosinophil count of <=6/HPF across all esophageal levels at the final treatment period evaluation. Participant was considered as responder at Week 16 if he/she achieved a minimum of 30% reduction in DSQ combined score between baseline and Week 16 and has peak eosinophil count of <=6/HPF across all esophagus levels. Number of participants with overall binary response I after 12 weeks of double blind treatment at Week 16 were reported.
Time Frame: Week 16
Population: FAS included all randomized participants who received at least one dose of a double-blind IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 105 | 213
Participants
  Overall Binary Response I: Responders | 0 | 64
  Overall Binary Response I: Non Responders | 105 | 149
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); Overall binary response I at the final treatment period was performed based on firth logistic regression model adjusted for age group and diet restriction; Test type: Superiority; p = 0.001, Firth logistic regression; Odds Ratio (OR) = 91.86, 95% CI 2-sided [5.687 to 1483.680]

10. Secondary Outcome: Number of Participants With Overall Binary Response II at the Final Treatment Period Evaluation (Week 16)
Description: Overall binary response II was defined as a reduction in the DSQ score of >=50% from baseline to the final treatment period evaluation and a peak eosinophil count of <=6/HPF across all esophageal levels at the final treatment period evaluation. Participant was considered as responder at Week 16 if he/she achieved a minimum of 50% reduction in DSQ combined score between baseline and Week 16 and had peak eosinophil count of <=6/HPF across all esophagus levels. Number of participants with overall binary response II after 12 weeks of double blind treatment at Week 16 were reported.
Time Frame: Week 16
Population: FAS included all randomized participants who received at least one dose of a double-blind IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 105 | 213
Participants
  Overall binary response II: Responders | 0 | 48
  Overall binary response II: Non-Responders | 105 | 165
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); Overall binary response II at the final treatment period was perfomed based on based on firth logistic regression model adjusted for age group and diet restriction; Test type: Superiority; p = 0.004, Firth logistic regression; Odds Ratio (OR) = 61.68, 95% CI 2-sided [3.836 to 991.858]

11. Secondary Outcome: Change From Baseline in the Dysphagia Symptom Questionnaire (DSQ) + Pain Score (Questions 2 +3+4) at the Final Treatment Period Evaluation (Week 16)
Description: DSQ contained 4 questions, all participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). DSQ + pain score was calculated by summing the scores of responses to questions 2, 3, and 4 by using following formula: DSQ + pain score= ([sum of points from questions 2+3+4 in the daily DSQ] ×14)/ Number of diaries reported with non-missing data. Scale range was 0 - 2 for question 2, 0 - 4 for question 3 and 0 - 4 for question 4, with higher values representing a worse outcome. Scale range for DSQ + pain score was 0 - 140, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 89 | 197
Score on scale | -12.24 (2.097) | -18.65 (1.660)
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); This analysis was from the analysis of covariance (ANCOVA) model with treatment group and age group as factors and the baseline DSQ + Pain score as a continuous covariate; Test type: Superiority; p = 0.004, ANCOVA; Difference in Least square mean = -6.41, 95% CI [-10.757 to -2.063]

12. Secondary Outcome: Change From Baseline in the Dysphagia Symptom Questionnaire (DSQ) Pain Score (Question 4) at the Final Treatment Period Evaluation (Week 16)
Description: DSQ pain score was calculated by summing the scores of responses to Question 4 (extent to which the participant experienced pain while swallowing) only, by using the following formula: DSQ pain score= [(sum of points from question 4 in the daily DSQ)×14]/ Number of diaries reported with non-missing data. Scale range was 0 - 4 for question 4, with higher values representing a worse outcome. Scale range for DSQ pain score was 0 - 56, with higher values representing a worse outcome. A negative change from baseline indicates that symptoms decreased. Change from baseline in DSQ pain score (question 4) after 12 weeks of double blind treatment at Week 16 were reported.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 89 | 197
score on scale | -3.01 (0.751) | -5.47 (0.595)
Statistical Analysis 1: Comparison: Placebo vs Oral Budesonide Suspension (OBS); This analysis was from the analysis of covariance (ANCOVA) model with treatment group and age group as factors and the baseline DSQ Pain score as a continuous covariate; Test type: Superiority; p = 0.002, ANCOVA; Difference in Least square mean = -2.46, 95% CI [-4.018 to -0.909]

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AE)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs that start or deteriorate on or after the first dose of double-blind IP (Week 44) and through the safety follow-up contact, or 31 days after the last dose of IP for participants who did not have a safety follow-up contact. Number of participants with TEAE's were reported.
Time Frame: From start of study drug administration up to follow-up (Week 20)
Population: Safety analysis set included all participants who received at least one dose of any double-blind IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 105 | 213
Participants | 64 | 130

14. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUCtau) Between the Defined Interval of Budesonide Doses
Description: Area under the curve for the defined interval between doses (12 hours), calculated using the linear-up/log-down trapezoidal rule.The AUCtau of plasma budesonide was reported. Hours times pico grams per milliliter was abbreviated as h.pg/mL.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Week 8, 12 and 16
Population: PK set included all participants in the safety set who received BOS treatment and provided at least one quantifiable plasma concentration of budesonide. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.pg/mL
Arm/Group | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 24
h.pg/mL | 5071 (58.1)

15. Secondary Outcome: Maximum Observed Concentration (Cmax) of Budesonide in Plasma
Description: The Cmax of budesonide in plasma was reported.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Week 8, 12 and 16
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter (pg/mL)
Arm/Group | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 47
Picograms per milliliter (pg/mL) | 914.8 (59.2)

16. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Budesonide in Plasma
Description: Tmax of budesonide in plasma was reported.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Week 8, 12 and 16
Population: as for outcome 14
Measure: Median (Full Range); unit: hour
Arm/Group | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 47
hour | 2 [0.50 to 4]

17. Secondary Outcome: Terminal Rate Constant (Lambda Z) of Budesonide in Plasma
Description: Lambda Z of budesonide in plasma was reported.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Week 8, 12 and 16
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 23
per hour | 0.2103 (25.2)

18. Secondary Outcome: Terminal Half-Life (t1/2) of Budesonide in Plasma
Description: t1/2 of budesonide in plasma was reported
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Week 8, 12 and 16
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 23
hour | 3.296 (25.2)

19. Secondary Outcome: Apparent Oral Clearance (CL/F) of Budesonide in Plasma
Description: CL/F of budesonide in plasma was reported.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Week 8, 12 and 16
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 24
Liter per hour (L/h) | 394.4 (58.1)

20. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Budesonide in Plasma
Description: Vz/F of budesonide in plasma was reported.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 12 hours post-dose on Week 8, 12 and 16
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Oral Budesonide Suspension (OBS)
Number analyzed (Participants) | 23
Liter (L) | 1886 (51.4)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Week 20)
Arm/Group | Placebo | Oral Budesonide Suspension (OBS)
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/213
Serious Adverse Events (participants affected / at risk) | 1/105 | 2/213
Other Adverse Events (participants affected / at risk) | 28/105 | 63/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=105) | Oral Budesonide Suspension (OBS) (N=213)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=105) | Oral Budesonide Suspension (OBS) (N=213)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (6)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (6) | 4 (4)
Nasopharyngitis (Infections and infestations) | 4 (6) | 11 (13)
Oesophageal candidiasis (Infections and infestations) | 2 (2) | 8 (8)
Oral candidiasis (Infections and infestations) | 0 (0) | 8 (9)
Sinusitis (Infections and infestations) | 3 (3) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (5)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
ACTH stimulation test abnormal (Investigations) | 3 (3) | 6 (7)
Protein urine present (Investigations) | 3 (4) | 1 (1)
Urine leukocyte esterase positive (Investigations) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 7 (7)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (5)
Mood swings (Psychiatric disorders) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Acne (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT02605837/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT02605837/SAP_001.pdf